CLINICAL TRIAL: NCT02610634
Title: Visual Function During Gait in Parkinson's Disease: Impact of Cognition and Response to Visual Cues
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: 6601; CLRN (Other: 125425); REC number (Other: 13/NE/0128)
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Older adults; Vision; Cognition; Visual cues; Eye-tracking; Gait; Saccades; Dual task; Visual sampling
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's disease: People with Parkinson's disease (≥ 50 years old) who do not have dementia (MoCA ≥ 21).
- Older Adults: Aged-matched older adults (≥ 50 years old) who are cognitively intact (MoCA ≥26).

SUMMARY:
Parkinson's disease (PD) is associated with problems of gait such as veering, difficulty turning, an inability to perceive doorways or obstacles, and negotiate uneven terrain. Gait problems, especially veering, may be exacerbated by visuospatial dysfunction which predispose to falls, freezing and festination of gait. Visuospatial dysfunction is common in PD and likely involves peripheral features (e.g. contrast sensitivity) as well as central cognitive mechanisms (e.g. attention).

Central neuro-degeneration in PD, PD dementia, and dementia with Lewy Bodies may influence visual function, as impaired visual sampling has been reported in these conditions. Visual sampling is measured via saccadic (fast eye movement) activity, as saccades are the mechanisms through which people orientate and explore the environment. The use of objective devices to reliably measure saccades is important to detect disease related eye movement changes. Emerging visuomotor research has measured visual sampling in PD using devices such as electrooculography and infra-red eye tracking, revealing reduced amplitude, speed and frequency of saccades during various tasks.

Despite recent increases in visuomotor research it remains unclear how PD influences visual sampling of the environment during gait and the influence of attentional and cognitive deficits. Recent work demonstrated that people with PD sample their environment less frequently than controls, despite a slower gait. Saccadic timing was unchanged in response to environmental cues. Despite this, environmental visual cues (transverse lines on the floor) have been shown to increase the number of fixations made during gait. However the mechanisms of this response remain unclear. Cognition is likely of importance, with response potentially influenced by attentional control.

This observational study aims to examine the influence of cognition on visuomotor control during gait in PD. This aim will be achieved by observation of visual sampling under several environmental challenges (straight walk, doorways, turns, visual cue) and a dual task.

DETAILED DESCRIPTION:
This is an observational study of visual sampling during gait under different environmental challenge (straight, doorway, turn and visual cue (transverse lines on the floor)) and dual task. These conditions represent everyday activities/environments which can be difficult for people with PD.

This is not an interventional study as participants are not assigned to any specific interventions by the researchers, or followed up to re-assess outcomes other than for reliability testing of the eye-tracking devices used. The study has been ethically approved (NRES Committee North East - Newcastle & North Tyneside 1: 13/NE/0128) as an observational study as participants are assigned to pre-defined groups, and have behavioural measures (primarily visual sampling and secondly gait) observed in the gait laboratory under various walking conditions common to everyday environments.

Study Hypotheses

The over-arching hypothesis of this observational study is that visual sampling during gait in PD will be influenced by cognitive impairments. This study hypothesises that saccadic activity will be restricted in PD compared to controls during gait. Dual task and environmental challenge via a doorway, turn or visual cue will influence saccadic activity during gait.

Specific study hypothesises are:

1. Cognition will selectively impact on visuomotor control during gait
2. Visual sampling strategies during gait will be related to selected domains of cognitive impairment

Secondary questions include:

1. Is the Dikablis mobile eye-tracker a reliable means of measuring saccadic activity in PD and healthy controls?

After undergoing screening to confirm eligibility, subjects will be assigned into one of two groups:

1. Older adult controls (HC; up to n = 40)
2. People with PD (n = 60)

   Recruitment

   Participants will be recruited from Movement Disorder Clinics in Newcastle upon-Tyne. Research personnel will be available at clinics as required to invite participants to consider the study. If sufficiently interested, participants will be given a Participant Information Sheet (PIS) and letter concerning the study. The invitation will be followed up by a telephone call during the week to assess willingness to participate. If willing, a mutually convenient time for assessment will be organised, and the invitation to attend will be extended to a carer or spouse.

   The healthy control group will be recruited via advertisement using posters, which will be placed within neurology and geriatric departments. The advertisement will also be sent via the university email system to staff and students at Newcastle University, the recipients will be advised to pass on the poster to potential interested parties (i.e. family or friends). All participants will be evaluated at the Clinical Ageing Research Unit, Newcastle University, a purpose-build research facility.

   Testing Protocol

   Session 1; (up to 150min)
   * Initial screening and baseline assessments (45-60min)
   * Visual sampling during gait (60-90min)

   Session 2; (up to 60min)

   • 1st Reliability testing (45-60min) (if applicable; for a subgroup of PD and HC participants)

   Session 3; (up to 60min)

   • 2nd Reliability testing (45-60min) (if applicable; for a subgroup of PD and HC participants)

   Visual sampling during gait (session 1)

   Participants (n=100) will be assessed in the gait laboratory at the clinical ageing and research unit (CARU), where they will walk under different conditions, for example single task, dual task, through a doorway, whilst turning and with a visual cue (transverse lines on the floor 50cm apart) in place. Visual sampling will be assessed with a Dikablis head-mounted eye tracking and electrooculography (EOG) systems. Gait will be simultaneously assessed using a 3D motion capture system (Vicon), which will be synchronised with the eye tracking systems to provide simultaneous data collection. Infra-red markers will be taped to the body and limbs of the subjects using a small amount of double-sided tape, to allow for motion tracking. The Dikablis will also be taped to the forehead of each participant using a small amount of double sided tape.

   Reliability testing (subgroup) (session 2 and 3)

   In order to examine the test re-test reliability of mobile eye-tracking in people with PD and healthy controls, a subgroup of participants (PD and HC; up to n=25) will return for a second (within approx. 1 week) and third visit. They will be asked to repeat some of the walking tasks outlined above and to sit (with chin rest), stand and walk (on a treadmill) while performing several eye movements to visual targets (horizontal and vertical visual angles such as; 5, 10, 15, 20 degrees) in time with an auditory cue (a 60bpm metronome). Participants will return for the third visit approx. 1 week after the second visit and repeat the reliability testing (as above).

   Sample Size

   This is an exploratory study and therefore few specific previous examples are available to guide the sample size required. The sample size estimate is based on results from previous work in this research area (PD; n=21) (Galna et al., 2012), other previous similar studies and preliminary pilot work with the Dikabilis mobile eye-tracker, which is a new instrument. Similar studies in this research area have used similar sample sizes (n=2-26), demonstrating that differences between PD and HC groups will been evident.

   Statistical Analysis

   Analysis Common to all Studies

   Statistical analysis will be undertaken using SPSS version 19 or more recent versions (SPPS, Inc. an IBM company). Data checks of all data collected will be carried out independently by two members of the Human Movement Science Team at the Clinical Ageing Research Unit to ensure that data is accurate.

   All statistical tests will be carried out at the 5% two-sided level of significance. Demographic characteristics and baseline data will be summarized using descriptive statistics, including means, standard deviations, median, minimum, maximum and inter-quartile ranges for continuous or ordinal data and percentages for categorical data. The descriptive statistics will be tabulated and presented graphically for clarity.The assessments recorded at pre-testing will be taken as baseline values.

   One-sample Kolmogorov-Smirnov tests will be used to check for normally distributed data. Non-normally distributed continuous distributions will be transformed where appropriate to meet the requirements of parametric tests; otherwise equivalent non-parametric tests will be adopted.

   Further Analysis

   To analyse visual sampling during gait Pearson's correlations will be used to test the strength and direction of the relationships between clinical, gait and saccadic outcomes. Analysis of variance (ANOVA) will be used to analyse the effect of group (PD, HC), dual task (single task, dual task) and environmental challenge (Straight walk, Door, Turn, Visual cue) on visual sampling during gait.

   To analyse reliability repeated-measure t-tests, Bland and Altman plots, intra-class correlation coefficients (Model 2, 1) and Pearson correlations (or non-parametric equivalents) will be used to assess bias, agreement and consistency of saccadic outcomes measured with the Dikablis eye-tracker on two separate occasions a week apart.

ELIGIBILITY:
Inclusion Criteria:

Common to all groups

* Aged ≥50 years
* Able to walk unaided
* Adequate hearing (as evaluated by the whisper test; stand 2m behind participant and whisper a 2 syllable word, participant repeats word) and vision capabilities (as measured using a Snellen chart - 6/18-6/12).
* Stable medication for the past 1 month and anticipated over a period of 6 months

Group Specific Criteria

Participants with PD:

* Diagnosis of idiopathic PD, as defined by the UK Brain Bank criteria
* Hoehn and Yahr stage I-III
* Stable medication for past 1 month and anticipated over next 6 months or stable Deep Brain Stimulation for at least one month and expected following 6 months
* Score ≥21/30 on Montreal cognitive assessment (MoCA) which is used to classify non-demented PD (PD dementia is <21/30)
* Free from any neurological disorders that may have caused cognitive impairment
* No restriction was made for medication usage and participants on stable doses of medication or treatment were permitted.

Exclusion Criteria:

Common to all groups

* Psychiatric co-morbidity (e.g., major depressive disorder as determined by geriatric depression scale (GDS-15); >10/15)
* Clinical diagnosis of dementia or other severe cognitive impairment (PD = MoCA <21/30, Controls = MoCA <26/30)
* History of stroke, traumatic brain injury or other neurological disorders (other than PD, for that group)
* Acute lower back or lower extremity pain, peripheral neuropathy, rheumatic and orthopaedic diseases
* Unstable medical condition including cardio-vascular instability in the past 6 months
* Unable to comply with the testing protocol or currently participating in another interfering research project
* Interfering therapy

Vision specific Criteria

* Any pupillary diameter disorder; such as significantly non-round pupils, Adies pupil (tonic or dilated pupil), Argyll-Robertson pupil (absence of light reaction), unilateral small pupil
* Neuromotility disorders, such as Nystagmus or other ocular oscillations
* Significant left eye disorders (i.e. squint, twitching, Ptosis [drooping eyelids])
* Known significant visual field deficits; such as hemianopia
* Optic nerve disease
* Optic disc elevation
* Optic disc swelling; such as Papilledema or Papillitis

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease participants will be recruited from Movement Disorder Clinics in Newcastle upon-Tyne.
  Healthy control older adults will be recruited locally within the Newcastle upon Tyne region.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Rochester, PhD, Principal Investigator — Newcastle University
Locations (1):
- Clinical Ageing Research Unit, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Background] Lord S, Galna B, Coleman S, Yarnall A, Burn D, Rochester L. Cognition and gait show a selective pattern of association dominated by phenotype in incident Parkinson's disease. Front Aging Neurosci. 2014 Oct 21;6:249. doi: 10.3389/fnagi.2014.00249. eCollection 2014. PMID 25374538
- [Background] Galna B, Lord S, Daud D, Archibald N, Burn D, Rochester L. Visual sampling during walking in people with Parkinson's disease and the influence of environment and dual-task. Brain Res. 2012 Sep 14;1473:35-43. doi: 10.1016/j.brainres.2012.07.017. Epub 2012 Jul 20. PMID 22824332
- [Result] Stuart S, Alcock L, Galna B, Lord S, Rochester L. The measurement of visual sampling during real-world activity in Parkinson's disease and healthy controls: a structured literature review. J Neurosci Methods. 2014 Jan 30;222:175-88. doi: 10.1016/j.jneumeth.2013.11.018. Epub 2013 Nov 27. PMID 24291711
- [Result] Stuart S, Galna B, Lord S, Rochester L, Godfrey A. Quantifying saccades while walking: validity of a novel velocity-based algorithm for mobile eye tracking. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:5739-42. doi: 10.1109/EMBC.2014.6944931. PMID 25571299
- [Result] Stuart S, Hickey A, Galna B, Lord S, Rochester L, Godfrey A. iTrack: instrumented mobile electrooculography (EOG) eye-tracking in older adults and Parkinson's disease. Physiol Meas. 2017 Jan;38(1):N16-N31. doi: 10.1088/1361-6579/38/1/N16. Epub 2016 Dec 12. PMID 27941232
- [Result] Stuart S, Lord S, Hill E, Rochester L. Gait in Parkinson's disease: A visuo-cognitive challenge. Neurosci Biobehav Rev. 2016 Mar;62:76-88. doi: 10.1016/j.neubiorev.2016.01.002. Epub 2016 Jan 7. PMID 26773722
- [Result] Stuart S, Galna B, Lord S, Rochester L. A protocol to examine vision and gait in Parkinson's disease: impact of cognition and response to visual cues. F1000Res. 2015 Nov 30;4:1379. doi: 10.12688/f1000research.7320.2. eCollection 2015. PMID 27092242

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Parkinson's Disease | Older Adults
Started | 60 | 40
Completed | 60 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parkinson's Disease | Older Adults | Total
Number analyzed (Participants) | 60 | 40 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (7.6) | 66.9 (10.9) | 67.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 38 | 23 | 61
Region of Enrollment [Number; unit: participants]
  United Kingdom | 60 | 40 | 100

OUTCOME MEASURES:

1. Primary Outcome: Visual Sampling Parameter: Saccade Frequency During Gait
Description: Number of fast eye movements made per second observed when walking, measured via EOG and Dikablis mobile eye-tracker. Walking conditions include; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins)
Measure: Mean (Standard Deviation); unit: Saccade frequency (sacc/sec)
Arm/Group | Parkinson's Disease | Older Adults
Number analyzed (Participants) | 56 | 40
Saccade frequency (sacc/sec)
  Straight Walk single task | 0.48 (0.54) | 0.76 (0.62)
  Straight Walk with Door single task | 0.67 (0.61) | 0.77 (0.57)
  Left Turn with Door single task | 1.05 (0.54) | 1.31 (0.60)
  Right Turn with Door single task | 1.01 (0.65) | 1.17 (0.74)
  Straight Walk dual task | 0.31 (0.37) | 0.53 (0.49)
  Straight Walk with Door dual task | 0.39 (0.39) | 0.60 (0.42)
  Left Turn with Door dual task | 0.81 (0.53) | 1.18 (0.61)
  Right Turn with Door dual task | 0.69 (0.51) | 1.11 (0.66)

2. Secondary Outcome: Gait Parameter: Gait Speed
Description: Measured in meters per second observed when walking recorded via Vicon 3D motion capture. Walking conditions include; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins)
Reporting Status: Not Posted

3. Secondary Outcome: Gait Parameter: Step Length
Description: Measured in meters recorded via Vicon 3D motion capture. Observed during the following walking conditions; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins)
Reporting Status: Not Posted

4. Secondary Outcome: Gait Parameter: Step Time
Description: Measured in seconds recorded via Vicon 3D motion capture. Observed during the following walking conditions; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins) and one week later in Session 2 for a sub-group (PD and controls n = upto 25) (lasting approx. 60mins)
Reporting Status: Not Posted

5. Secondary Outcome: Gait Parameter: Single Support Time
Description: as for outcome 4
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins)
Reporting Status: Not Posted

6. Secondary Outcome: Gait Parameter: Double Support Time
Description: as for outcome 4
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins)
Reporting Status: Not Posted

7. Secondary Outcome: Visual Sampling Parameter: Saccade Number During Gait
Description: Number of fast eye movements observed when walking, measured via EOG and Dikablis mobile eye-tracker. Walking conditions include; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: as for outcome 4
Reporting Status: Not Posted

8. Secondary Outcome: Visual Sampling Parameter: Saccade Velocity During Gait
Description: Velocity (degrees per second) of fast eye movements observed when walking, measured via EOG and Dikablis mobile eye-tracker. Walking conditions include; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins)
Reporting Status: Not Posted

9. Secondary Outcome: Visual Sampling Parameter: Saccade Amplitude During Gait
Description: Distance (degrees) of fast eye movements observed when walking, measured via EOG and Dikablis mobile eye-tracker. Walking conditions include; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins)
Reporting Status: Not Posted

10. Secondary Outcome: Visual Sampling Parameter: Saccade Acceleration During Gait
Description: Acceleration (degrees per second squared) of fast eye movements observed when walking, measured via EOG and Dikablis mobile eye-tracker. Walking conditions include; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins)
Reporting Status: Not Posted

11. Secondary Outcome: Visual Sampling Parameter: Fixation Number During Gait
Description: Number of pauses (fixations) between fast eye movements observed when walking, measured via EOG and Dikablis mobile eye-tracker. Walking conditions include; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins)
Reporting Status: Not Posted

12. Secondary Outcome: Visual Sampling Parameter: Fixation Duration During Gait
Description: Duration (ms) of pauses (fixations) between fast eye movements observed when walking, measured via EOG and Dikablis mobile eye-tracker. Walking conditions include; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins)
Reporting Status: Not Posted

13. Secondary Outcome: Visual Sampling Parameter: Saccade Duration During Gait
Description: Duration (ms) of fast eye movements observed when walking, measured via EOG and Dikablis mobile eye-tracker. Walking conditions include; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: Session 1: observation during gait assessments (lasting approx. 90mins)
Reporting Status: Not Posted

14. Secondary Outcome: Visual Sampling Parameter: Number of Blinks During Gait
Description: Number of blinks observed when walking, measured via EOG and Dikablis mobile eye-tracker. Walking conditions include; single task, dual task, through a doorway, whilst turning and with a visual cue in place.
Time Frame: as for outcome 4
Reporting Status: Not Posted

15. Other Pre Specified Outcome: CDR Attention Battery (Cognitive Drug Research - CDR, United Biosource Corporation, UK)
Description: The Attention CDR involves a series of computerised tests, which the subjects respond to by pressing one of two buttons. Scores for sub-sections of Simple reaction time, Digit vigilance and Choice reaction time will be obtained.
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Benton's Judgement of Line Orientation (JLO) Test
Description: JLO is a test of visuospatial ability, which involves a subject viewing a set of numbered lines and then being shown two lines of the same orientation. Participants then have to name the numbers that the shown lines correspond to.
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Clock Copying (CLOX 1 and 2)
Description: Participants are required to draw a clock with the numbers and arrows pointed at a particular time. Then the subjects have to copy a clock drawn by the researcher.
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Visual Object and Space Perception Battery (VOSP)
Description: This study will use a selection of these tests; incomplete letters, dot counting and position discrimination.
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Visual Acuity
Description: VA is measured binocularly used a standard LogMAR chart. Participants will be seated at a distance of 4m from the chart. Participants will be instructed to read aloud down the chart starting from the top left.
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Contrast Sensitivity
Description: CS will be measured using the Mars CS sheets placed on an adjustable holder. The sheet consists of 48 Latin letters of uniform height; the contrast from the white background decreases with subsequent letters. Room illumination is adjusted so that average CS sheet luminance is between 80 and 120cd/m² (measured via a luminance meter). Assessment is done binocularly with the average distance from the patients eyes being 50cm. Participants read aloud down the sheet starting at the top left. Errors are recorded on the pre-set score sheet and testing is terminated after 2 consecutive errors.
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

21. Other Pre Specified Outcome: The Unified Parkinson's Disease Rating Scale (UPDRS)
Description: The Unified Parkinson's Disease Rating Scale will be used to assess motor and non-motor features of PD and disease severity. The UPDRS is scored from a total of 195 points; higher scores reflect worsening disability.
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Hoehn & Yahr (H & Y) Scale
Description: The Hoehn and Yahr rating scale is a widely used clinical rating scale, which defines broad categories of motor function in Parkinson's disease (PD). All participants' will be tested who are in H &Y stages I-III.
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Freezing of Gait (FOG) Questionnaire
Description: This is a 10 item questionnaire intended to classify freezing of gait. The questionnaire has 3 parts; distinction of freezers from non-freezers, Freezing severity, frequency and duration and impact of freezing on daily life.
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Falls Efficacy Scale - International (FES-I)
Description: Fear of falling will be measured using the falls efficacy scale - international version. This is a short and valid measure of fear of falling in older adults, which assesses basic and demanding activities (both physical and social). It consists of 16 scenarios (e.g. cleaning the house) and subjects must rate their fear of falling on a scale from 1 (Not at all concerned) to 4 (Very concerned).
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Montreal Cognitive Assessment (MoCA)
Description: Different cognitive domains are assessed (attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation).
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Addenbrookes Cognitive Examination (ACE-R)
Description: The ACE-R involves testing of attention, orientation, memory, fluency, language and visuospatial abilities.
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Geriatric Depression Scale (GDS-15)
Description: This involves 15 questions about the mood of the subjects. Scores of 0 to 4 to be in the normal range, 5 to 9 to indicate mild depression, and 10 to 15 to indicate moderate to severe depression.
Time Frame: Session 1 (full session lasts approx. 3 hours)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Parkinson's Disease | Older Adults
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/40
Other Adverse Events (participants affected / at risk) | 0/60 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No